CLINICAL TRIAL: NCT01849731
Title: Effectiveness of Two Interventions in Patients With Low Educational Level With Diabetes to Reduce Inequalities in Self-care Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andalusian School of Public Health (Other Government)
Responsible Party: Principal Investigator, Clara Bermúdez-Tamayo, PhD in Health Economics, Andalusian School of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI-0096-2010
Record Dates: First submitted 2013-05-06; First posted 2013-05-08 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Diabetes Mellitus type 2;; Primary Care, healthcare inequalities;; Diabetes self-management,; Quality of diabetes care
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention A (Experimental): Face-to face intervention
  Interventions: Other: Face-to-face
- Intervention B (Experimental): Face-to-face intervention plus telephone reinforcement
  Interventions: Other: Face-to-face intervention plus telephone reinforcement
- Control Group (No Intervention)

INTERVENTIONS:
Other: Face-to-face — is carried out by the GPs during the clinic visit and consists of seven visits, one every three months. Each session consists of completing a diabetes care record sheet (DCRS) together with the patient. The DCRS consists of two parts: Five questions on self-care activities in the last three months and a graph with previously measured HbA1c levels. This information is completed at each session, resulting in a graph showing the evolution of glycaemic control related to self-care activities. The DCRS is explained patients, emphasising the relationship between self-care and glycemic control. At the end of the session, patients are given a copy of the DCRS and suggested to show it and discuss it with their relatives.
  Arms: Intervention A
Other: Face-to-face intervention plus telephone reinforcement — In this group patients receive the above described intervention A plus a telephone reinforcement It consists on five telephone calls lasting about 10 minutes each, to provide advice on carrying out physical exercise and eating a balanced diet and to encourage the use of health services related to diabetes control. Any problems or doubts that patients have stemming from any aspect of diabetes care are also discussed. Telephone reinforcement is carried out by a professional who has previously been trained in promoting T2DM self-management and in motivational interviewing techniques.
  Arms: Intervention B

SUMMARY:
The purpose of this cluster randomized trial is to determine whether an intervention implemented in a General Surgery, based in improving patient-provider communication, results in a better diabetes self-management in patients with lower educational level. A secondary objective is to assess whether telephone reinforcement enhances the effect of such intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DM2,
* Over 18 years,
* Low educational level (no college to GBS or ESO),
* Inadequate glycemic control (glycosylated hemoglobin levels above 7%)

Exclusion Criteria:

* Physical or mental condition that prevents the completion of the intervention - complications arising from severe DM2 altering routine medical monitoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2011-02; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Glycosylated Haemoglobin levels | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Andalussian School of Public Health, Granada, Granada, Spain

REFERENCES:
- [Derived] Ricci-Cabello I, Olry de Labry-Lima A, Bolivar-Munoz J, Pastor-Moreno G, Bermudez-Tamayo C, Ruiz-Perez I, Quesada-Jimenez F, Moratalla-Lopez E, Dominguez-Martin S, de los Rios-Alvarez AM, Cruz-Vela P, Prados-Quel MA, Lopez-De Hierro JA. Effectiveness of two interventions based on improving patient-practitioner communication on diabetes self-management in patients with low educational level: study protocol of a clustered randomized trial in primary care. BMC Health Serv Res. 2013 Oct 23;13:433. doi: 10.1186/1472-6963-13-433. PMID 24153053